CLINICAL TRIAL: NCT02264678
Title: A Modular Phase I, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumour Activity of Ceralasertib in Combination With Cytotoxic Chemotherapy and/or DNA Damage Repair/Novel Anti-cancer Agents in Patients With Advanced Solid Malignancies.
Brief Title: Ascending Doses of Ceralasertib in Combination With Chemotherapy and/or Novel Anti Cancer Agents
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5330C00004; 2023-505006-41-00 (Registry Identifier: CTIS (EU)); 2014-002233-66 (EudraCT Number)
Expanded Access: NCT03079687 (Approved for marketing)
Record Dates: First submitted 2014-07-30; First posted 2014-10-15 (Estimated); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Adv Solid Malig - H&N SCC, ATM Pro / Def NSCLC, Gastric, Breast and Ovarian Cancer
Keywords: ATM deficient, ATM proficient, HER2 negative, Breast, Gastric, Head & Neck, Lung, Ovarian
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib; durvalumab; AZD5305; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Module 2 Part A1 (Experimental): Module 2 Part A1: ascending doses of ceralasertib will be administered alone to define the maximum tolerated dose (MTD) and/or a continuous, tolerable Recommended Dose (RD) to take into Module 2 Part A2.
  Interventions: Drug: Administration of ceralasertib
- Module 2 Part A2 (Experimental): Module 2 Part A2: ascending doses of ceralasertib will be administered in combination with olaparib to patients to define the dose, frequency and schedule of ceralasertib and olaparib to take into Module 2 Part B.
  Interventions: Drug: Administration of ceralasertib in combination with olaparib
- Module 2 Part B1 (Experimental): Module 2 Part B1: Patients with second line 'ATM deficient' gastric adenocarcinoma including GEJ adenocarcinoma will receive ceralasertib with olaparib, at dose, frequency and schedule recommended from Module 2 Part A2.
  Interventions: Drug: Administration of ceralasertib in combination with olaparib
- Module 2 Part B2 (Experimental): Module 2 part B2: Patients with second line 'ATM proficient' gastric adenocarcinoma including GEJ adenocarcinoma will receive ceralasertib with olaparib, at dose, frequency and schedule recommended from Module 2 Part A2.
  Interventions: Drug: Administration of ceralasertib in combination with olaparib
- Module 2 Part B3 (Experimental): Module 2 Part B3: Patient with second or third line breast cancer with BRCA mutations (somatic or germline), excluding HER2 positive breast cancer will receive ceralasertib with olaparib, at dose, frequency and schedule recommended from Module 2 Part A2.
  Interventions: Drug: Administration of ceralasertib in combination with olaparib
- Module 2 Part B4 (Experimental): Module Part B4: Patients with second or third line triple negative breast cancer with no known BRCA mutations. This expansion will be enriched for patients with disease harbouring a HRR-related gene mutation (HRRm) will receive ceralasertib with olaparib, at dose, frequency and schedule recommended from Module 2 Part A2.
  Interventions: Drug: Administration of ceralasertib in combination with olaparib
- Module 3 Part A (Experimental): Module 3 Part A: cohort escalation of ceralasertib in combination with durvalumab in HNSCC or NSCLC patients to define the dose, frequency and schedule of ceralasertib and durvalumab to take into Module 3 Part B. Additionally, Module 3 Part A will include a serial tumour biopsy cohort to evaluate the Proof of Mechanism of ceralasertib in HNSCC and NSCLC patients.
  Interventions: Drug: Administation of ceralasertib in combination with durvalumab
- Module 3 Part B (Experimental): Module 3 Part B: cohort expansions of ceralasertib in combination with durvalumab in HNSCC or NSCLC patients at dose, frequency and schedule from Module 3 Part A.
  Interventions: Drug: Administation of ceralasertib in combination with durvalumab
- Module 2 Part B5 (Experimental): Patients with BRCA mutant or RAD51C/D mutant (either germline or somatic) or HRD-positive status epithelial ovarian, fallopian tube, or primary peritoneal cancer according to local testing. Patients must be platinum sensitive and previously progressed on a licensed PARPi. The cohort will be split into 2 groups: Cohort 1 - without intervening chemotherapy following progression on a PARPi, Cohort 2 - with intervening chemotherapy following progression on a PARPi. Patients will receive ceralasertib and olaparib, at the RP2D dose, frequency and schedule established from Module 2 Part A2.
  Interventions: Drug: Administration of ceralasertib in combination with olaparib
- Module 4 (FE/QT) (Experimental): Ceralasertib monotherapy will be administered on a number of days during Cycle 0 to assess the effect of food on ceralasertib absorption and effect of ceralasertib on ECG parameters under various conditions (fasted, fed, steady state). From C1 onwards, patients who participated in C0 will be allocated to either ceralasertib in combination with olaparib or durvalumab, or ceralasertib monotherapy and assessed for safety.
  Interventions: Drug: Administration of ceralasertib monotherapy; Drug: Administration of ceralasertib and olaparib; Drug: Administration of ceralasertib and durvalumab
- Module 5 Part A (Experimental): Module 5 Part A: ascending doses of ceralasertib will be administered in combination with AZD5305 to patients to define the MTD, RP2D.
  In case this first dose level is not tolerated, alternative schedules will be evaluated.
  Interventions: Drug: Administration of ceralasertib in combination with AZD5305
- Module 5 Part B (Experimental): Module 5 Part B: cohort expansions of ceralasertib in combination with AZD5305 in ovarian patients at dose, frequency and schedule from Module 5 Part A.
  Interventions: Drug: Administration of ceralasertib in combination with AZD5305
- Module 1 Part A (Experimental): Module 1 Part A: ascending doses of ceralasertib in combination with carboplatin AUC5 will be administered to patients to define the maximum tolerated dose (MTD) and/or a continuous, tolerable Recommended Dose (RD).
  Interventions: Drug: Administration of ceralasertib in combination with carboplatin
- Module 1 Part B (Experimental): Module 1 Part B: patients with advanced lung adenocarcinoma with low expression of ATM will receive ceralasertib and carboplatin, at the dose, frequency and schedule recommended from Module 1 Part A.
  Interventions: Drug: Administration of ceralasertib in combination with carboplatin

INTERVENTIONS:
Drug: Administration of ceralasertib — An oral formulation of ceralasertib will be used. In Module 2 Part A1, patients will receive a single dose of ceralasertib on Day 1, followed by 4 to 6 days washout, before multiple dosing.
  Arms: Module 2 Part A1
Drug: Administration of ceralasertib in combination with olaparib — An oral formulations of ceralasertib and olaparib will be used. In Module 2 Part A2, patients will receive either a single or twice daily dose of ceralasertib followed by 4 to 6 days washout, before multiple dosing with ceralasertib and olaparib. In Module 2 Part B, patients will receive ceralasertib and olaparib at the dose, frequency and schedule recommended from Module 2 Part A2. Cycle 0 may be omitted at the discretion of the sponsor.
  Arms: Module 2 Part A2; Module 2 Part B1; Module 2 Part B2; Module 2 Part B3; Module 2 Part B4; Module 2 Part B5
Drug: Administation of ceralasertib in combination with durvalumab — An oral formulation of ceralasertib will be used. Durvalumab is given via IV infusion. In Module 3 Part A, patients will receive an initial single dose of ceralasertib on Day 1, followed by multiple dosing in combination with durvalumab. In Module 3 Serial Tumour Biopsy Extension and Part B expansion cohorts, patients will receive ceralasertib at the dose, frequency and schedule recommended from Module 3 Part A, in combination with durvalumab.
  Arms: Module 3 Part A; Module 3 Part B
Drug: Administration of ceralasertib monotherapy — Module 4 Part A and Module 4 Part B Cohort 3: During C0, patients will receive ceralasertib monotherapy orally once a day on 3 non-consecutive days and ceralasertib twice a day on 5 consecutive days. After the patients have completed C0 (Part A) they may transition to Module 4 Part B cohort 3 where they will continue to receive ceralasertib monotherapy
  Arms: Module 4 (FE/QT)
Drug: Administration of ceralasertib and olaparib — Module 4 Part B Cohort 1:
  After completion of Part A (C0), the patient may transition to Part B and be allocated to receive ceralasertib in combination with olaparib as decided by the investigator.
  Arms: Module 4 (FE/QT)
Drug: Administration of ceralasertib and durvalumab — Module 4 Part B Cohort 2:
  After completion of Part A (C0), the patient may transition to Part B and be allocated to receive ceralasertib in combination with durvalumab as decided by the investigator.
  Arms: Module 4 (FE/QT)
Drug: Administration of ceralasertib in combination with AZD5305 — An oral formulations of ceralasertib and AZD5305 will be used. In Module 5 Part A, patients will receive a single dose of ceralasertib on cycle 0 Day 1 as per dose level cohort. In Module 5 Part B, patients will receive ceralasertib and AZD5305: C1 onwards (as per dose level cohort allocated).
  Arms: Module 5 Part A; Module 5 Part B
Drug: Administration of ceralasertib in combination with carboplatin — An oral formulation of ceralasertib will be used. In Module 1 Part A, patients will receive a single dose of ceralasertib on Day 1, followed by multiple dosing in combination with carboplatin. A maximum of 6 cycles (21 days per cycle) of treatment will be given. In Module 1 Part B, patients will receive ceralasertib and carboplatin at the dose, frequency and schedule recommended from Module 1 Part A.
  Arms: Module 1 Part A; Module 1 Part B

SUMMARY:
This is a modular, phase I/ phase 1 b, open-label, multicentre study of ceralasertib administered orally in combination with cytotoxic chemotherapy regimens and/or novel anti-cancer agents, to patients with advanced malignancies. The study design allows an investigation of optimal combination dose of ceralasertib with other anti-cancer treatments, with intensive safety monitoring to ensure the safety of the patients. The initial combination to be investigated is ceralasertib with carboplatin. The second combination to be investigated is ceralasertib with Olaparib. The third combination to be investigated is ceralasertib with durvalumab. The fourth module will investigate the effect of food on ceralasertib absorption and the effect of ceralasertib on ECG parameter. The fifth module to be investigated is ceralasertib with AZD5305.

DETAILED DESCRIPTION:
This is a modular, phase I, two part, open-label, multicentre study of ceralasertib, administered orally, in combination with cytotoxic chemotherapy regimens and/or novel anti-cancer agents, to patients with advanced/metastatic solid malignancies. The study design allows an escalation of the dose of ceralasertib in combination with the standard dose and schedule of either cytotoxic chemotherapies and/or novel anti-cancer agents, with intensive safety monitoring to ensure the safety of the patients. There are two parts to each combination module of this study; part A, dose escalation and an optional part B, cohort expansions in particular patient groups. The initial combination module will be with Carboplatin (module 1). The second combination will be with Olaparib (module 2). The third combination will be with durvalumab (module 3), the fourth combination will be AZD5305 (Module 5). The option to start further combination modules will be the decision of the Safety Review Committee (SRC), based on emerging preclinical data and, safety and tolerability information from the initial combination. Combinations of ceralasertib with novel anti-cancer agents may also be explored. Once a minimally biologically active dose of ceralasertib, for that combination module, has been identified from part A of that module, the SRC may decide to commence part B if deemed to be necessary. This may include cohort expansions of specific patient groups to explore preliminary anti-tumour activity or the effect of food or particular drug combinations on drug pharmacokinetics. The fourth module will investigate the effect of food on ceralasertib absorption and whether ceralasertib has an effect on QT.

ELIGIBILITY:
Principal Inclusion criteria:

* Aged at least 18
* The presence of a solid malignant tumour that is not considered appropriate for further standard treatment
* Module 2 Part B study expansions, and Module 3: patients must have a tumour at least 1 cm in size that can be measured using a CT or MRI scan
* Module 2 Part B All (except B5): No previous treatment with PARP inhibitor.
* Module 2 Part B1 Study expansion: advanced gastric adenocarcinoma (including GEJ) patients with ATM deficient tumours
* Module 2 Part B2 Study expansion: advanced gastric adenocarcinoma (including GEJ) patients with ATM proficient tumours
* Module 2 Part B3 Study expansion: Second or thrid line HER2 negative breast cancer
* Module 2 Part B4 Study expansion: Second or third line triple negative breast cancer (TNBC)
* Module 2 Part B5 Study expansion: BRCAm or RAD51C/Dm or PALB2m or HRD positive status ovarian cancer patient who are Platinum Sensitive Relapsed and have previously progressed on a licensed PARPi
* Module 3: advanced recurrent or metastatic non-small cell lung cancer, or head and neck squamous cell carcinoma
* Module 4: any advanced solid tumours except gastric, gastro-oesophageal, oesophageal or colorectal cancer with a small bowel resection
* Module 4: Ability to comply with an overnight fast of at least 10 hours prior to dosing and 4 hours after dosing as mandated, and ability to eat a high fat meal as mandated
* Module 5 All: Ovarian fallopian tube or primary peritonial cancer, previous treatment with PARP inhibitor, platinum-sensitive relapsed ovarian cancer
* Module 5 Part B: known or suspected BRCA mutation, PALB2 mutation, RAD51C/D mutation or HRD positive status

Principal exclusion criteria

* A diagnosis of ataxia telangiectasia
* Prior exposure to an ATR inhibitor
* Bad reaction to ceralasertib
* Module 2: Contra-indicated for treatment with olaparib
* Module 3: Contra-indicated for treatment with durvalumab
* Module 4: Mean resting corrected QT interval (QTc) >470 msec or history of familial long QT syndrome.
* Module 4: Patients with type I or type II diabetes
* Module 5: Known hypersensitivity to PARP including AZD5305

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of subjects with adverse events/serious adverse events | From baseline until 28 days after discontinuation of study treatment for Module 1, 2 and 5 or until 90 days after discontinuation of study treatment for Module 3 and 4
  Number of patients with adverse events and with serious adverse events including abnormal clinical observations, DLT, abnormal Electrocardiogram (ECG) parameters, abnormal laboratory assessments and abnormal vital signs that changed from baseline.
Module 4 only: Effect of food on ceralasertib absorption by Intensive PK assessments after a single oral dose of ceralasertib (Part A) | From 0h to 24h on Day 2 and Day15 in Cycle 0 (Part A) - Cycle 0 is 15 days
  Intensive PK sampling at defined timepoints to measure Geometric mean and 90% CI for the ratio of fed:
  fasted in area under the plasma concentration time curve from zero to the last measurable time point (AUC0-t), area under the plasma concentration time curve from zero to infinity (AUC)
Module 4 only: Effect of ceralasertib on ECG parameters (HR, PR, QRS and QTcF) by ECG recordings | From 0h to 24h on Day 2, Day 8 and Day15 in Cycle 0 (Part A) - Cycle 0 is 15 days
  Change from baseline HR, PR, QRS and QTcF (ΔHR, ΔPR, ΔQRS and ΔQTcF) Categorical outliers for QTcF, HR, PR, and QRS Frequency of treatment emergent T and U wave abnormalities If a substantial HR effect is observed (i.e., the absolute value of the largest least squares [LS] mean ΔHR is greater than 10bpm in the by-time point analysis), other correction methods such as individualised and optimised individualised HR corrected QT interval (QTcI) will be explored and compared.
  The method that removes the HR dependence of the QT interval most efficiently will be chosen as the primary correction method.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of ceralasertib | At predefined intervals throughout the ceralasertib treatment period (approximately 8 weeks for Module 1 and 16 weeks + IP disc. for Module 2+3)
  Blood samples will be collected to assess plasma concentration of ceralasertib at a series of time points to derive Cmax.
Time to observed Cmax (Tmax) for ceralasertib | At predefined intervals throughout the ceralasertib treatment period (approximately 8 weeks for Module 1 and 16 weeks + IP disc. for Module 2+3)
  Blood samples will be collected to assess plasma concentration of ceralasertib at a series of time points to derive Tmax.
Area under the plasma concentration-time curve (AUC) for ceralasertib | At predefined intervals throughout the ceralasertib treatment period (approximately 8 weeks for Module 1 and 16 weeks + IP disc. for Module 2+3)
  Blood samples will be collected to assess plasma concentration of ceralasertib at a series of time points to derive AUC.
Maximum Observed Plasma Concentration (Cmax) of Carboplatin | At predefined intervals throughout the Carboplatin treatment period (approximately 4 weeks for Module 1)
  Blood samples will be collected to assess plasma concentration of Carboplatin at a series of time points to derive Cmax.
Time to observed Cmax (Tmax) for Carboplatin | At predefined intervals throughout the Carboplatin treatment period (approximately 4 weeks for Module 1)
  Blood samples will be collected to assess plasma concentration of Carboplatin at a series of time points to derive Tmax.
Area under the plasma concentration-time curve (AUC) for Carboplatin | At predefined intervals throughout the Carboplatin treatment period (approximately 4 weeks for Module 1)
  Blood samples will be collected to assess plasma concentration of Carboplatin at a series of time points to derive AUC.
Maximum Observed Plasma Concentration (Cmax) of Olaparib | At predefined intervals throughout the Olaparib treatment period (approximately 12 weeks for Module 2)
  Blood samples will be collected to assess plasma concentration of Olaparib at a series of time points to derive Cmax.
Time to observed Cmax (Tmax) for Olaparib | At predefined intervals throughout the Olaparib treatment period (approximately 12 weeks for Module 2)
  Blood samples will be collected to assess plasma concentration of Olaparib at a series of time points to derive Tmax.
Area under the plasma concentration-time curve (AUC) for Olaparib | At predefined intervals throughout the Olaparib treatment period (approximately 12 weeks for Module 2)
  Blood samples will be collected to assess plasma concentration of Olaparib at a series of time points to derive AUC.
Maximum Observed Plasma Concentration (Cmax) of durvalumab | At predefined intervals throughout the durvalumab treatment period (approximately 28 weeks + 90days post IP disc. for Module 3)
  Blood samples will be collected to assess plasma concentration of durvalumab at a series of time points to derive Cmax.
Time to observed Cmax (Tmax) for durvalumab | At predefined intervals throughout the durvalumab treatment period (approximately 28 weeks + 90days post IP disc. for Module 3)
  Blood samples will be collected to assess plasma concentration of durvalumab at a series of time points to derive Tmax.
Area under the plasma concentration-time curve (AUC) for durvalumab | At predefined intervals throughout the durvalumab treatment period (approximately 28 weeks + 90days post IP disc. for Module 3)
  Blood samples will be collected to assess plasma concentration of durvalumab at a series of time points to derive AUC.
Assessment of pharmacodynamic biomarker changes | Biopsies of tumour at baseline and last day of dosing
  Evaluation of ceralasertib activity in the tumour by assessment of pharmacodynamic biomarker changes which may include, but are not limited to functional ATR inhibition, ctDNA and CTCs.
Best objective response | From first dose to confirmed progressive disease (approximately 1 year)
  Best objective response will be determined for each patient based on the best response recorded from start of study treatment to end of treatment, including any assessments for confirmation after the end of treatment using RECIST 1.1.
Objective response rate | From first dose to confirmed progressive disease (approximately 1 year)
  Objective response rate is defined as the percentage of patients who have at least one response of CR or PR prior to any evidence of progression (as defined by RECIST 1.1) that is confirmed at least 4 weeks later.
Percentage change in tumour size | From first dose to confirmed progressive disease (approximately 1 year)
  Percentage change in tumour size will be determined for patients with measurable disease at baseline and is derived at each visit by the percentage change from baseline in the sum of the diameters of TLs. The best percentage change in tumour size will be the patient's value representing the largest decrease (or smallest increase) from baseline in tumour size using RECIST 1.1.
Durable response rate | From first documented response to confirmed progressive disease (approximately 1 year)
  Duration of response will be defined as the time from the date of first documented response until date of documented progression or death in the absence of disease progression, the end of response should coincide with the date of progression or death from any cause used for the PFS endpoint using RECIST 1.1.
Progression free survival | From first dose to confirmed progressive disease (approximately 1 year)
  Progression free survival (PFS) is defined as the time from start of treatment (first dose of ceralasertib) until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the subject withdraws from therapy or receives another anti-cancer therapy prior to progression using RECIST 1.1.
Survival assessment /status | From first dose to confirmed progressive disease (approximately 1 year)
  Module 2 only. To be obtained for all patients who received ceralasertib and olaparib in part A2, B1, B2, B3, B4 and B5.
Module 4: Safety and tolerability in terms of AE and SAE as recorded in safety measures | From baseline until 28 days after discontinuation of study treatment for Module 4 Part B cohort 1 and cohort 3, or until 90 days after discontinuation of study treatment for Module 4 Part B cohort 2
  Safety measures: AEs assessments (CTCAE grading)
Module 4 only: Effect of food on ceralasertib absorption by Cmax in a fasted and fed state (Part A) | Part A (Cycle 0 Day 2/Day 8/Day 15) - each cycle is of 15 days
  Intensive PK sampling at defined timepoints to measure geometric mean and 90% CI for the ratio of fed: fasted in Cmax - Maximum plasma concentration (Cmax)
Module 4 only: Effect of food on ceralasertib absorption by Tmax in a fasted and fed state (Part A) | Part A (Cycle 0 Day 2/Day 8/Day 15) - each cycle is of 15 days
  Intensive PK sampling at defined timepoints to measure geometric mean and 90% CI for the ratio of fed: fasted in Tmax - time to reach maximum plasma concentration (Tmax)
Module 4 only: Effect of food on ceralasertib absorption by clearance in a fasted and fed state (Part A) | Part A (Cycle 0 Day 2/Day 8/Day 15) - each cycle is of 15 days
  Intensive PK sampling at defined timepoints to measure geometric mean and 90% CI for the ratio of fed: fasted in apparent clearance following oral administration (CL/F)
Module 4 only: Effect of food on ceralasertib absorption by apparent volume of distribution in a fasted and fed state (Part A) | Part A (Cycle 0 Day 2/Day 8/Day 15) - each cycle is of 15 days
  Intensive PK sampling at defined timepoints to measure geometric mean and 90% CI for the ratio of fed: fasted in apparent volume of distribution (Vz/F)
Module 4 only: Effect of food on ceralasertib absorption by terminal half-life and terminal rate constant in a fasted and fed state (Part A) | Part A (Cycle 0 Day 2/Day 8/Day 15) - each cycle is of 15 days
  Intensive PK sampling at defined timepoints to measure geometric mean and 90% CI for the ratio of fed: fasted in terminal rate constant (λz), and terminal half-life (t1/2)
Module 4: The number of subjects with adverse events/serious adverse events | From baseline until 28 days after discontinuation of study treatment for Module 4 Part B cohort 1 and cohort 3, or until 90 days after discontinuation of study treatment for Module 4 Part B cohort 2
  Number of patients with adverse events and with serious adverse events including abnormal clinical observations, abnormal vital signs, and abnormal laboratory assessments that changed from baseline
Module 5 only: Maximum Observed Plasma Concentration (Cmax) of AZD5305 | At predefined intervals throughout AZD5305 treatment period (approximately 8 weeks + IP disc)
  Blood samples will be collected to assess plasma concentration of AZD5305 at a series of time points to derive Cmax.
Module 5 only: Time to observed Cmax (Tmax) for AZD5305 | At predefined intervals throughout AZD5305 treatment period (approximately 8 weeks + IP disc)
  Blood samples will be collected to assess plasma concentration of AZD5305 at a series of time points to derive Tmax.
Module 5 only: Area under the plasma concentration-time curve (AUC) for AZD5305 | At predefined intervals throughout AZD5305 treatment period (approximately 8 weeks + IP disc)
  Blood samples will be collected to assess plasma concentration of AZD5305 at a series of time points to derive AUC.

CONTACTS AND LOCATIONS:
Locations (22):
- United States (7):
  - Research Site, Duarte, California
  - Research Site, Irvine, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York
  - Research Site, Philadelphia, Pennsylvania
- France (4):
  - Research Site, Bordeaux
  - Research Site, Lyon
  - Research Site, Saint-Herblain
  - Research Site, Villejuif
- South Korea (3):
  - Research Site, Goyang-si
  - Research Site, Seongnam-si
  - Research Site, Seoul
- United Kingdom (8):
  - Research Site, Bristol
  - Research Site, Cambridge
  - Research Site, Coventry
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Oxford
  - Research Site, Sutton
  - Research Site, Withington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Smith G, Alholm Z, Coleman RL, Monk BJ. DNA Damage Repair Inhibitors-Combination Therapies. Cancer J. 2021 Nov-Dec 01;27(6):501-505. doi: 10.1097/PPO.0000000000000561. PMID 34904813